CLINICAL TRIAL: NCT02675426
Title: A Phase 3, Randomized, Double-Blind Study Comparing Upadacitinib (ABT-494) to Placebo in Subjects With Moderately to Severely Active Rheumatoid Arthritis Who Are on a Stable Dose of Conventional Synthetic Disease-Modifying Anti-Rheumatic Drugs (csDMARDs) and Have an Inadequate Response to csDMARDs
Brief Title: A Study Comparing Upadacitinib (ABT-494) to Placebo in Adults With Rheumatoid Arthritis on a Stable Dose of Conventional Synthetic Disease-Modifying Antirheumatic Drugs (csDMARDs) Who Have an Inadequate Response to csDMARDs Alone
Acronym: SELECT-NEXT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-549; 2015-003332-13 (EudraCT Number)
Record Dates: First submitted 2015-12-11; First posted 2016-02-05 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Musculoskeletal Disease; Arthritis; Joint Disease; Anti-inflammatory agents; Antirheumatic agents; Upadacitinib; ABT-494
MeSH Terms: conditions — Arthritis, Rheumatoid; Musculoskeletal Diseases; Arthritis; Joint Diseases | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Upadacitinib 15 mg (Experimental): Period 1: Participants receive upadacitinib 15 mg once daily for 12 weeks.
  Period 2: Participants continue to receive upadacitinib 15 mg once daily for an additional 248 weeks.
  Interventions: Drug: Upadacitinib
- Upadacitinib 30 mg (Experimental): Period 1: Participants receive upadacitinib 30 mg once daily for 12 weeks.
  Period 2: Participants continue to receive upadacitinib 30 mg once daily for an additional 248 weeks or until implementation of Protocol Amendment 6 at which time participants switch to receive upadacitinib 15 mg once daily.
  Interventions: Drug: Upadacitinib
- Placebo / Upadacitinib 15 mg (Experimental): Period 1: Participants receive placebo once daily for 12 weeks.
  Period 2: Participants receive upadacitinib 15 mg once daily for 248 weeks.
  Interventions: Drug: Placebo; Drug: Upadacitinib
- Placebo / Upadacitinib 30 mg (Experimental): Period 1: Participants receive placebo once daily for 12 weeks.
  Period 2: Participants receive upadacitinib 30 mg once daily for 248 weeks or until implementation of Protocol Amendment 6 at which time participants switch to receive upadacitinib 15 mg once daily.
  Interventions: Drug: Placebo; Drug: Upadacitinib

INTERVENTIONS:
Drug: Placebo — Tablet; Oral
  Arms: Placebo / Upadacitinib 15 mg; Placebo / Upadacitinib 30 mg
Drug: Upadacitinib — Tablet; Oral
  Other Names: ABT-494; Rinvoq

SUMMARY:
The primary objectives of this study are to compare the efficacy, safety, and tolerability of upadacitinib 30 mg once daily (QD) and 15 mg QD versus placebo for the treatment of signs and symptoms of adults with moderately to severely active rheumatoid arthritis who were on a stable dose of csDMARDs and had an inadequate response to csDMARDs.

DETAILED DESCRIPTION:
This Phase 3 multicenter study includes two periods. Period 1 is a 12-week, randomized, double-blind, parallel-group, placebo-controlled period designed to compare the safety and efficacy of upadacitinib 30 mg once daily and upadacitinib 15 mg once daily versus placebo for the treatment of signs and symptoms of adults with moderately to severely active rheumatoid arthritis (RA) who were on a stable dose of csDMARDs and had an inadequate response to csDMARDs.

Period 2 is a 248-week blinded long-term extension period to evaluate the long-term safety, tolerability, and efficacy of upadacitinib 30 mg once daily and upadacitinib 15 mg once daily in participants who completed Period 1.

Participants were to be randomized in a 2:2:1:1 ratio using interactive response technology (IRT) to receive double-blind study drug in one of the following treatment groups:

* Group 1: Upadacitinib 30 mg QD in Period 1 → Upadacitinib 30 mg QD in Period 2
* Group 2: Upadacitinib 15 mg QD in Period 1 → Upadacitinib 15 mg QD in Period 2
* Group 3: Placebo in Period 1 → Upadacitinib 30 mg QD in Period 2
* Group 4: Placebo in Period 1 → Upadacitinib 15 mg QD in Period 2

Randomization was stratified by prior exposure to biological disease-modifying anti-rheumatic drug (bDMARD) (yes/no) and geographic region.

Following Protocol Amendment 6.0 approval in December 2019, all participants still on study received open-label upadacitinib 15 mg QD, including those on upadacitinib 30 mg QD, with the earliest switch occurring at the Week 168 visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, at least 18 years old.
* Diagnosis of rheumatoid arthritis (RA) for greater than or equal to 3 months.
* Subjects have been receiving conventional synthetic DMARD (csDMARD) therapy for greater than or equal to 3 months and on a stable dose for greater than or equal to 4 weeks prior to the first dose of study drug. The following csDMARDs are allowed: methotrexate (MTX), sulfasalazine, hydroxychloroquine, chloroquine, and leflunomide.
* Meets the following minimum disease activity criteria: greater than or equal to 6 swollen joints (based on 66 joint counts) and greater than or equal to 6 tender joints (based on 68 joint counts) at Screening and Baseline Visits.
* Subjects with prior exposure to at most one biologic DMARD (bDMARD) may be enrolled (up to 20% of study population) if they have documented evidence of intolerance to bDMARDs or limited exposure (less than 3 months) and have satisfied required washout periods.

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor (including but not limited to tofacitinib, baricitinib, and filgotinib).
* History of inflammatory joint disease other than RA. History of secondary Sjogren's Syndrome is permitted.
* Subjects who are considered inadequate responders to bDMARD therapy as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (167):
- United States (57):
  - AZ Arthritis and Rheum Assoc /ID# 148651, Mesa, Arizona
  - SunValley Arthritis Center, Lt /ID# 140452, Peoria, Arizona
  - AZ Arthritis and Rheum Researc /ID# 138500, Phoenix, Arizona
  - AZ Arthritis and Rheum Researc /ID# 139286, Phoenix, Arizona
  - AZ Arthritis & Rheuma Research /ID# 138598, Phoenix, Arizona
  - Arizona Research Center, Inc. /ID# 140448, Phoenix, Arizona
  - University of Arizona Cancer Center - North Campus /ID# 140451, Tucson, Arizona
  - Covina Arthritis Clinic /ID# 139881, Covina, California
  - T. Joseph Raoof, MD, Inc. /ID# 140964, Encino, California
  - Allergy and Rheum Med Clin /ID# 146082, La Jolla, California
  - Pacific Arthritis Ctr Med Grp /ID# 138744, Los Angeles, California
  - Robin K. Dore MD, Inc /ID# 138688, Tustin, California
  - Inland Rheum Clin Trials Inc. /ID# 138853, Upland, California
  - Denver Arthritis Clinic /ID# 139876, Denver, Colorado
  - Clinical Res of West FL, Inc. /ID# 138854, Clearwater, Florida
  - Ctr Arthritis & Rheumatic Dise /ID# 141696, Miami, Florida
  - Medallion Clinical Research Institute, LLC /ID# 140074, Naples, Florida
  - Suncoast Clinical Research /ID# 138633, New Port Richey, Florida
  - Omega Research Consultants /ID# 139877, Orlando, Florida
  - Arthritis Center, Inc. /ID# 141363, Palm Harbor, Florida
  - Institute of Arthritis Res /ID# 138548, Idaho Falls, Idaho
  - OrthoIllinois /ID# 139695, Rockford, Illinois
  - Clinical Investigation Special /ID# 139696, Skokie, Illinois
  - Springfield Clinic /ID# 138602, Springfield, Illinois
  - Deerbrook Medical Associates /ID# 139694, Vernon Hills, Illinois
  - Indiana Univ School of Med /ID# 140077, Indianapolis, Indiana
  - Bluegrass Community Research /ID# 138295, Lexington, Kentucky
  - Four Rivers Clinical Research /ID# 141134, Paducah, Kentucky
  - MMP Women's Health /ID# 141542, Portland, Maine
  - The Center for Rheumatology & /ID# 139203, Wheaton, Maryland
  - Mansfield Health Center /ID# 141357, Mansfield, Massachusetts
  - Advanced Rheumatology, PC /ID# 140071, Lansing, Michigan
  - Justus J. Fiechtner, MD, PC /ID# 138697, Lansing, Michigan
  - Physician Res. Collaboration /ID# 138533, Lincoln, Nebraska
  - Westroads Clinical Research /ID# 138304, Omaha, Nebraska
  - The Center for Rheumatology /ID# 138746, Albany, New York
  - PMG Research of Salisbury /ID# 141023, Salisbury, North Carolina
  - PMG Research of Wilmington LLC /ID# 140951, Wilmington, North Carolina
  - Cincinnati Rheumatic Disease Study Group, Inc. /ID# 138868, Cincinnati, Ohio
  - Arthritis Assoc of NW Ohio /ID# 140953, Toledo, Ohio
  - Health Research Oklahoma /ID# 138535, Oklahoma City, Oklahoma
  - Altoona Ctr Clinical Res /ID# 138741, Duncansville, Pennsylvania
  - Articularis Healthcare Group, Inc d/b/a Low Country Rheumatology /ID# 138689, Summerville, South Carolina
  - Comprehensive Arthritis Care, a division of Comprehensive Rheumatology Care PLLC /ID# 141021, Hendersonville, Tennessee
  - Tekton Research, Inc. /ID# 141428, Austin, Texas
  - Trinity Universal Res Assoc /ID# 149271, Carrollton, Texas
  - Arth and Osteo Clin Brazo Valley /ID# 147809, College Station, Texas
  - Metroplex Clinical Research /ID# 138698, Dallas, Texas
  - Baylor College of Medicine /ID# 138682, Houston, Texas
  - Houston Institute for Clin Res /ID# 138716, Houston, Texas
  - Arthritis Consultants, P.A. /ID# 141138, Killeen, Texas
  - Trinity Universal Research Association /ID# 148649, Plano, Texas
  - Accurate Clinical Management /ID# 139338, San Antonio, Texas
  - Arthritis & Osteoporosis Clinic /ID# 138703, Waco, Texas
  - Western Washington Arthritis C /ID# 138728, Bothell, Washington
  - Arthritis Northwest, PLLC /ID# 138539, Spokane, Washington
  - Aurora Rheumatology and Immunotherapy Center /ID# 139306, Franklin, Wisconsin
- Argentina (2):
  - Mautalen Salud e Investigacion /ID# 141419, Buenos Aires
  - Inst. Rheumatologic Strusberg /ID# 145648, Córdoba
- Australia (4):
  - Coffs Clinical Trials /ID# 138747, Coffs Harbour, New South Wales
  - Optimus Clinical Research Pty. /ID# 138769, Kogarah, New South Wales
  - Emeritus Research /ID# 138773, Camberwell, Victoria
  - Barwon Rheumatology /ID# 138772, Geelong, Victoria
- Austria (2):
  - Rheuma Zentrum Favoriten GmbH /ID# 138787, Vienna
  - Wilhelminenspital der Stadt Wien /ID# 138788, Vienna
- Belgium (3):
  - Rhumaconsult SPRL /ID# 138813, Charleroi, Hainaut
  - UZ Gent /ID# 138806, Ghent, Oost-Vlaanderen
  - AZ Sint Lucas /ID# 141338, Bruges
- Bosnia and Herzegovina (2):
  - University Clinical Centre of the Republic of Srpska /ID# 138819, Banja Luka, Republika Srpska
  - University Clinical Centre of the Republic of Srpska /ID# 140372, Banja Luka, Republika Srpska
- Bulgaria (2):
  - Diag Consult Ctr 17 Sofia EOOD /ID# 141006, Sofia
  - Diagnostic Consultative Center /ID# 138882, Sofia
- Canada (4):
  - Manitoba Clinic /ID# 139086, Winnipeg, Manitoba
  - Eastern Health /ID# 140431, St. John's, Newfoundland and Labrador
  - Groupe de Recherche en Maladies Osseuses /ID# 138906, Sainte-Foy, Quebec
  - Dr. Latha Naik /ID# 139089, Saskatoon, Saskatchewan
- Croatia (4):
  - Klinicki bolnicki centar Rijeka /ID# 138649, Rijeka, Primorje-Gorski Kotar County
  - Klinicka bolnica Sveti Duh /ID# 152812, Zagreb
  - Medical Center Kuna-Peric /ID# 140365, Zagreb
  - Poliklinika Bonifarm /ID# 141415, Zagreb
- Czechia (5):
  - L.K.N. Arthrocentrum, s.r.o /ID# 141340, Hlučín, Moravskoslezský kraj
  - Revmatologie, s.r.o. /ID# 138899, Brno
  - Artroscan s.r.o. /ID# 138833, Ostrava
  - Nemocnice Slany /ID# 141112, Slaný
  - PV-MEDICAL s.r.o. /ID# 138913, Zlín
- Estonia (3):
  - Center of Clinical and Basic Research /ID# 141116, Tallinn, Harju
  - Paernu Hospital /ID# 138961, Pärnu
  - East Tallinn Central Hospital /ID# 140618, Tallinn
- Finland (3):
  - Helsinki Univ Central Hospital /ID# 140381, Helsinki
  - Kiljava Medical Research /ID# 139260, Hyvinkää
  - South Karelia Central Hospital /ID# 139973, Lappeenranta
- France (2):
  - Hopital Saint Joseph /ID# 149188, Marseille, Bouches-du-Rhone
  - CHRU Tours - Hopital Trousseau /ID# 138969, Chambray-lès-Tours
- Germany (5):
  - Uniklinik Koln /ID# 139084, Cologne, North Rhine-Westphalia
  - Charité Universitätsmedizin Campus Mitte /ID# 139052, Berlin
  - Immanuel-Krankenhaus /ID# 139059, Berlin
  - Asklepios Klinik Altona /ID# 140466, Hamburg
  - Welcker, Planegg, DE /ID# 140467, Planegg
- University General Hospital of Heraklion "PA.G.N.I" /ID# 139115, Heraklion, Greece
- Prince of Wales Hospital /ID# 139314, Shatin, Hong Kong
- Hungary (2):
  - Revita Reumatologiai Rendelo /ID# 140761, Budapest
  - Fejer Megyei Szent Gyorgy Korh /ID# 138554, Székesfehérvár
- St Vincent's University Hosp /ID# 138562, Dublin, Ireland
- Universita di Catanzaro Magna Graecia /ID# 139316, Catanzaro, Calabria, Italy
- JSC Nat Scientific Med Res Ctr /ID# 140575, Astana, Kazakhstan
- LTD M+M Centers /ID# 138818, Ādaži, Latvia
- Lithuania (2):
  - Klaipeda University Hospital /ID# 141416, Klaipėda
  - Vilnius University Hospital /ID# 141348, Vilnius
- Mexico (2):
  - Centro Peninsular de Investigación Clínica SCP /ID# 148160, Colonia Centro, Yucatán
  - Unidad de Investigacion de las Enfermedades Reumatologicas SA de CV /ID# 138841, Mexico City
- Porter Rheumatology Ltd /ID# 138347, Nelson, New Zealand
- Poland (5):
  - NZOZ Nasz Lekarz /ID# 138374, Torun, Kuyavian-Pomeranian Voivodeship
  - McBk Sc /Id# 138360, Grodzisk Mazowiecki, Masovian Voivodeship
  - Osteo-Medic spolka cywilna /ID# 138371, Bialystok, Podlaskie Voivodeship
  - NZOZ Centrum Reumatologiczne /ID# 138353, Elblag, Warmian-Masurian Voivodeship
  - Rheuma Medicus /ID# 138372, Warsaw
- Portugal (2):
  - Instituto Portugues De Reumatologia /ID# 148315, Lisbon, Lisbon District
  - Centro Hospitalar Lisboa Ocidental, EPE /ID# 140594, Lisbon, Lisbon District
- School of Medicine University of Puerto Rico-Medical Sciences Campus /ID# 139328, San Juan, Puerto Rico
- Romania (3):
  - Spitalul Clinic Judetean de Urgenta /ID# 138407, Cluj-Napoca
  - Spitalul Municipal Ploiesti /ID# 138405, Ploieşti
  - Spitalul Clinic Judetean de Ur /ID# 138393, Sibiu
- Russia (7):
  - LLC Novaya Klinika /ID# 139269, Pyatigorsk, Stavropol Kray
  - Kazan State Medical University /ID# 138413, Kazan', Tatarstan, Respublika
  - Republican Clin Hos n.a. Baran /ID# 139273, Petrozavodsk
  - Samara Regional Clinical Hosp /ID# 148642, Samara
  - Ulyanovsk Regional Clin Hosp /ID# 139279, Ulyanovsk
  - Voronezh State Medical Univers /ID# 148431, Voronezh
  - Yaroslavi State Medical Univer /ID# 139908, Yaroslavl
- Slovakia (5):
  - ARTROMAC n.o. /ID# 138428, Košice
  - Nemocnica Kosice Saca, a.s. /ID# 138918, Košice
  - Slovak research center Team Member, Thermium s.r.o. /ID# 139924, Pieštany
  - Narodny ustav reumatickych chorob Piestany /ID# 138427, Pieštany
  - REUMA-GLOBAL, s.r.o. /ID# 139912, Trnava
- South Africa (3):
  - St. Augustine's Medical Centre /ID# 141352, Berea, KwaZulu-Natal
  - Arthritis Clinical Research Tr /ID# 138945, Cape Town, Western Cape
  - Winelands Medical Research Ctr /ID# 138944, Stellenbosch, Western Cape
- South Korea (9):
  - Inha University Hospital /ID# 149310, Incheon, Gwang Yeogsi
  - Ajou University Hospital /ID# 149311, Suwon, Gyeonggido
  - Chonnam National University Hospital /ID# 138651, Gwangju, Jeonranamdo
  - Hanyang University Seoul Hospi /ID# 138655, Seoul, Seongdong-gu
  - Cath Univ Seoul St Mary's Hosp /ID# 138652, Seoul, Seoul Teugbyeolsi
  - Daegu Catholic University Med /ID# 139249, Daegu
  - Chungnam National University Hospital /ID# 138653, Daejeon
  - Seoul National University Hospital /ID# 138659, Seoul
  - Asan Medical Center /ID# 140579, Seoul
- Spain (4):
  - Hospital Regional de Malaga /ID# 138975, Málaga, Malaga
  - Hospital General Univ de Elche /ID# 138991, Elche
  - Hospital Clin Univ San Carlos /ID# 138993, Madrid
  - Hosp Nuestra Senora Esperanza /ID# 138997, Santiago de Compostela
- HFR Fribourg - Hopital Canton /ID# 139155, Fribourg, Switzerland
- Taiwan (6):
  - China Medical University Hosp /ID# 139232, Taichung, Taichung
  - National Cheng Kung University Hospital /ID# 140868, Tainan, Tainan
  - National Taiwan Univ Hosp /ID# 141443, Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 140869, Kaohsiung City
  - Far Eastern Memorial Hospital /ID# 140871, New Taipei City
  - Taipei Veterans General Hosp /ID# 139234, Taipei
- Ankara Numune Training and Res /ID# 139237, Ankara, Turkey (Türkiye)
- Ukraine (3):
  - LLC Revmocentr /ID# 139872, Kyiv
  - MNCE "Lviv City Clinical Hospital #4" /ID# 139873, Lviv
  - Odessa National Medical Univ /ID# 139179, Odesa
- United Kingdom (6):
  - Leicester Royal Infirmary /ID# 139184, Leicester, England
  - Whipps Cross Univ Hospital /ID# 139523, London, London, City of
  - The Royal Free Hospital /ID# 139191, London, London, City of
  - Western General Hospital /ID# 139524, Edinburgh
  - Southampton General Hospital /ID# 139169, Southampton
  - Warrington + Halton Hosp NHS /ID# 139195, Warrington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Background] Burmester GR, Kremer JM, Van den Bosch F, Kivitz A, Bessette L, Li Y, Zhou Y, Othman AA, Pangan AL, Camp HS. Safety and efficacy of upadacitinib in patients with rheumatoid arthritis and inadequate response to conventional synthetic disease-modifying anti-rheumatic drugs (SELECT-NEXT): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2018 Jun 23;391(10139):2503-2512. doi: 10.1016/S0140-6736(18)31115-2. Epub 2018 Jun 18. PMID 29908669
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Burmester GR, Van den Bosch F, Tesser J, Shmagel A, Liu Y, Khan N, Camp HS, Kivitz A. Upadacitinib in Rheumatoid Arthritis and Inadequate Response to Conventional Synthetic Disease-Modifying Antirheumatic Drugs: Efficacy and Safety Through 5 Years (SELECT-NEXT). J Rheumatol. 2024 Jul 1;51(7):663-672. doi: 10.3899/jrheum.2023-1062. PMID 38621793
- [Derived] Rubbert-Roth A, Kakehasi AM, Takeuchi T, Schmalzing M, Palac H, Coombs D, Liu J, Anyanwu SI, Lippe R, Curtis JR. Malignancy in the Upadacitinib Clinical Trials for Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis. Rheumatol Ther. 2024 Feb;11(1):97-112. doi: 10.1007/s40744-023-00621-6. Epub 2023 Nov 20. PMID 37982966
- [Derived] Charles-Schoeman C, Choy E, McInnes IB, Mysler E, Nash P, Yamaoka K, Lippe R, Khan N, Shmagel AK, Palac H, Suboticki J, Curtis JR. MACE and VTE across upadacitinib clinical trial programmes in rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. RMD Open. 2023 Nov;9(4):e003392. doi: 10.1136/rmdopen-2023-003392. PMID 37945286
- [Derived] Fleischmann R, Curtis JR, Charles-Schoeman C, Mysler E, Yamaoka K, Richez C, Palac H, Dilley D, Liu J, Strengholt S, Burmester G. Safety profile of upadacitinib in patients at risk of cardiovascular disease: integrated post hoc analysis of the SELECT phase III rheumatoid arthritis clinical programme. Ann Rheum Dis. 2023 Sep;82(9):1130-1141. doi: 10.1136/ard-2023-223916. Epub 2023 Jun 12. PMID 37308218
- [Derived] Conaghan PG, Pavelka K, Hsieh SC, Bonnington TL, Kent TC, Marchbank K, Edwards CJ. Evaluating the efficacy of upadacitinib in patients with moderate rheumatoid arthritis: a post-hoc analysis of the SELECT phase 3 trials. Rheumatol Adv Pract. 2023 Feb 8;7(1):rkad017. doi: 10.1093/rap/rkad017. eCollection 2023. PMID 36794283
- [Derived] Burmester GR, Cohen SB, Winthrop KL, Nash P, Irvine AD, Deodhar A, Mysler E, Tanaka Y, Liu J, Lacerda AP, Palac H, Shaw T, Mease PJ, Guttman-Yassky E. Safety profile of upadacitinib over 15 000 patient-years across rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and atopic dermatitis. RMD Open. 2023 Feb;9(1):e002735. doi: 10.1136/rmdopen-2022-002735. PMID 36754548
- [Derived] Kakehasi AM, Radominski SC, Baravalle MD, Palazuelos FCI, Garcia-Garcia C, Arruda MS, Curi M, Liu J, Qiao M, Velez-Sanchez P, Vargas JI. Safety of upadacitinib in Latin American patients with rheumatoid arthritis: an integrated safety analysis of the SELECT phase 3 clinical program. Clin Rheumatol. 2023 May;42(5):1249-1258. doi: 10.1007/s10067-023-06513-y. Epub 2023 Jan 30. PMID 36715850
- [Derived] Bergman M, Buch MH, Tanaka Y, Citera G, Bahlas S, Wong E, Song Y, Zueger P, Ali M, Strand V. Routine Assessment of Patient Index Data 3 (RAPID3) in Patients with Rheumatoid Arthritis Treated with Long-Term Upadacitinib Therapy in Five Randomized Controlled Trials. Rheumatol Ther. 2022 Dec;9(6):1517-1529. doi: 10.1007/s40744-022-00483-4. Epub 2022 Sep 20. PMID 36125701
- [Derived] Bergman M, Tundia N, Yang M, Orvis E, Clewell J, Bensimon A. Economic Benefit from Improvements in Quality of Life with Upadacitinib: Comparisons with Tofacitinib and Methotrexate in Patients with Rheumatoid Arthritis. Adv Ther. 2021 Dec;38(12):5649-5661. doi: 10.1007/s12325-021-01930-4. Epub 2021 Oct 12. PMID 34636000
- [Derived] Yamaoka K, Tanaka Y, Kameda H, Khan N, Sasaki N, Harigai M, Song Y, Zhang Y, Takeuchi T. The Safety Profile of Upadacitinib in Patients with Rheumatoid Arthritis in Japan. Drug Saf. 2021 Jun;44(6):711-722. doi: 10.1007/s40264-021-01067-x. Epub 2021 May 27. PMID 34041702
- [Derived] Cohen SB, van Vollenhoven RF, Winthrop KL, Zerbini CAF, Tanaka Y, Bessette L, Zhang Y, Khan N, Hendrickson B, Enejosa JV, Burmester GR. Safety profile of upadacitinib in rheumatoid arthritis: integrated analysis from the SELECT phase III clinical programme. Ann Rheum Dis. 2021 Mar;80(3):304-311. doi: 10.1136/annrheumdis-2020-218510. Epub 2020 Oct 28. PMID 33115760
- [Derived] Strand V, Pope J, Tundia N, Friedman A, Camp HS, Pangan A, Ganguli A, Fuldeore M, Goldschmidt D, Schiff M. Upadacitinib improves patient-reported outcomes in patients with rheumatoid arthritis and inadequate response to conventional synthetic disease-modifying antirheumatic drugs: results from SELECT-NEXT. Arthritis Res Ther. 2019 Dec 9;21(1):272. doi: 10.1186/s13075-019-2037-1. PMID 31815649
- [Derived] Nader A, Mohamed MF, Winzenborg I, Doelger E, Noertersheuser P, Pangan AL, Othman AA. Exposure-Response Analyses of Upadacitinib Efficacy and Safety in Phase II and III Studies to Support Benefit-Risk Assessment in Rheumatoid Arthritis. Clin Pharmacol Ther. 2020 Apr;107(4):994-1003. doi: 10.1002/cpt.1671. Epub 2019 Nov 30. PMID 31610021
- See also: Related Info. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 149 centers in 35 countries in North America, eastern and western Europe, Asia, South America, Australia, New Zealand, and South Africa.
  The study included a 12-week placebo-controlled, double-blind period (Period 1), and a 5-year (248-week) double-blind extension (Period 2).
Pre-assignment Details: Participants were randomly assigned in a 1:1:2:2 ratio to one of the four treatment groups below. Randomization was stratified by prior exposure to biologic disease-modifying anti-rheumatic drug (bDMARD) and geographical region.
Groups:
- Placebo / Upadacitinib 15 mg: Participants received placebo once daily for 12 weeks in Period 1 followed by upadacitinib 15 mg once daily for 248 weeks in Period 2.
- Placebo / Upadacitinib 30 mg: Participants received placebo once daily for 12 weeks in Period 1 followed by upadacitinib 30 mg once daily for 248 weeks or until implementation of Protocol Amendment 6 at which time they were switched to receive upadacitinib 15 mg once daily.
- Upadacitinib 15 mg: Participants received upadacitinib 15 mg once daily for 12 weeks in Period 1 and continued to receive upadacitinib 15 mg once daily for an additional 248 weeks in Period 2.
- Upadacitinib 30 mg: Participants received upadacitinib 30 mg once daily for 12 weeks in Period 1. In Period 2 participants continued to receive upadacitinib 30 mg for an additional 248 weeks or until implementation of Protocol Amendment 6 at which time participants were switched to receive upadacitinib 15 mg once daily.
Period: Period 1: Week 1 to Week 12
Arm/Group | Placebo / Upadacitinib 15 mg | Placebo / Upadacitinib 30 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Started | 110 | 111 | 221 | 219
Received Study Drug | 110 | 111 | 221 | 219
Completed | 104 | 104 | 213 | 201
Not Completed | 6 | 7 | 8 | 18
Not completed — Adverse Event | 3 | 3 | 3 | 9
Not completed — Withdrawal by Subject | 1 | 2 | 5 | 5
Not completed — Lost to Follow-up | 0 | 1 | 0 | 2
Not completed — Other | 2 | 1 | 0 | 2
Period: Period 2: Week 12 to Week 260
Arm/Group | Placebo / Upadacitinib 15 mg | Placebo / Upadacitinib 30 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Started (Four participants completed the Week 12 visit but did not continue into Period 2.) | 103 | 103 | 212 | 200
Received Study Drug | 103 | 102 | 207 | 199
Switched to Upadacitinib 15 mg After Protocol Amendment 6 | 0 | 53 | 0 | 126
Completed | 61 | 49 | 130 | 120
Not Completed | 42 | 54 | 82 | 80
Not completed — Adverse Event | 13 | 16 | 17 | 30
Not completed — Withdrawal by Subject | 14 | 21 | 31 | 30
Not completed — Lost to Follow-up | 5 | 5 | 10 | 4
Not completed — Coronavirus Disease - 2019 (COVID-19) Infection | 1 | 0 | 0 | 1
Not completed — COVID-19 Logistic Restrictions | 1 | 0 | 1 | 0
Not completed — Other | 8 | 12 | 23 | 15

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) includes all randomized participants who received at least one dose of study drug.
  The two placebo groups are combined for analysis of results in Period 1.
Groups:
- Placebo: Participants randomized to receive placebo once daily for 12 weeks in Period 1.
- Upadacitinib 15 mg: Participants randomized to receive upadacitinib 15 mg once daily for 12 weeks in Period 1.
- Upadacitinib 30 mg: Participants randomized to receive upadacitinib 30 mg once daily for 12 weeks in Period 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg | Total
Number analyzed (Participants) | 221 | 221 | 219 | 661
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (12.22) | 55.3 (11.47) | 55.8 (11.29) | 55.7 (11.65)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 21 | 23 | 22 | 66
  40 to 64 years | 145 | 153 | 145 | 443
  ≥ 65 years | 55 | 45 | 52 | 152
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 182 | 172 | 520
  Male | 55 | 39 | 47 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 23 | 30 | 80
  Not Hispanic or Latino | 194 | 198 | 189 | 581
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 187 | 188 | 186 | 561
  Black or African American | 10 | 13 | 8 | 31
  American Indian / Alaskan Native | 1 | 0 | 1 | 2
  Asian | 19 | 19 | 21 | 59
  Multiple | 4 | 1 | 3 | 8
Geographical Region [Count of Participants; unit: Participants] — Other includes Australia, New Zealand, and South Africa.
  Participants
    North America | 90 | 88 | 89 | 267
    South/Central America | 8 | 10 | 11 | 29
    Western Europe | 24 | 22 | 23 | 69
    Eastern Europe | 74 | 76 | 73 | 223
    Asia | 16 | 17 | 15 | 48
    Other | 9 | 8 | 8 | 25
Prior Biological DMARD Use [Count of Participants; unit: Participants]
  Yes | 29 | 27 | 28 | 84
  No | 192 | 194 | 191 | 577
Duration of Rheumatoid Arthritis (RA) Diagnosis [Mean (Standard Deviation); unit: years] | 7.2 (7.45) | 7.3 (7.89) | 7.3 (7.86) | 7.3 (7.72)
Conventional Synthetic DMARD (csDMARD) Use at Baseline [Count of Participants; unit: Participants]
  Methotrexate alone | 141 | 122 | 136 | 399
  Methotrexate and other csDMARD | 49 | 47 | 39 | 135
  csDMARD other than methotrexate | 30 | 51 | 44 | 125
  Missing | 1 | 1 | 0 | 2
Tender Joint Count [Mean (Standard Deviation); unit: tender joints] — A total of 68 joints were assessed for the presence or absence of tenderness.
  tender joints | 24.7 (14.96) | 25.2 (13.80) | 26.2 (14.26) | 25.4 (14.34)
Swollen Joint Count [Mean (Standard Deviation); unit: swollen joints] — A total of 66 joints were assessed for the presence or absence of swelling.
  swollen joints | 15.4 (9.24) | 16.0 (10.04) | 16.2 (10.55) | 15.8 (9.95)
Patient's Assessment of Pain [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to indicate the severity of their arthritis pain within the previous week on a visual analog scale (VAS) from 0 to 100. A score of 0 indicates "no pain" and a score of 100 indicates "worst possible pain." Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 221 | 217 | 219 | 657
    (all) | 61.5 (20.80) | 64.1 (19.45) | 64.0 (19.77) | 63.2 (20.02)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: units on a scale] — The participant was asked to rate their current RA disease activity over the past 24 hours ranging from 0 to 100 using a VAS, where 0 indicates very low disease activity and 100 indicates very high disease activity. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 221 | 217 | 219 | 657
    (all) | 60.3 (20.50) | 63.1 (21.86) | 62.8 (20.32) | 62.1 (20.91)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: units on a scale] — The physician rated the participant's current global RA disease activity (independently from the participant's assessment) on a VAS scale from 0 to 100, where 0 indicates very low disease activity and 100 indicates very high disease activity. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 211 | 209 | 213 | 633
    (all) | 64.4 (17.67) | 64.3 (16.22) | 63.0 (17.99) | 63.9 (17.30)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 221 | 216 | 219 | 656
    (all) | 1.4 (0.63) | 1.5 (0.61) | 1.5 (0.61) | 1.5 (0.62)
High-sensitivity C-reactive Protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] | 12.6 (13.96) | 16.6 (19.17) | 14.8 (16.86) | 14.7 (16.86)
Disease Activity Score Based on CRP (DAS28 [CRP]) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A DAS28 score > 5.1 indicates high disease activity, a DAS28 score ≤ 3.2 indicates low disease activity, and a DAS28 score < 2.6 indicates clinical remission. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 221 | 217 | 219 | 657
    (all) | 5.6 (0.84) | 5.7 (0.97) | 5.7 (0.90) | 5.6 (0.91)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 12
Description: The primary endpoint for United States (US)/Food and Drug Administration (FDA) regulatory purposes was ACR 20% response (ACR20) at Week 12. Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity;
     * Patient global assessment of disease activity;
     * Patient assessment of pain;
     * Health Assessment Questionnaire - Disability Index (HAQ-DI);
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom ACR data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 221 | 221 | 219
percentage of participants | 35.7 [29.4 to 42.1] | 63.8 [57.5 to 70.1] | 66.2 [59.9 to 72.5]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — The overall type I error rate of the primary and ranked key secondary endpoints for the two doses was controlled using a graphical multiple testing procedure; p < 0.001, Cochran-Mantel-Haenszel — The adjusted p-value under multiplicity control is reported, with significance achieved if the adjusted p-value is less than 0.05; Cochran-Mantel-Haenszel test adjusted for the stratification factor of prior biological disease-modifying anti-rheumatoid drug use; Response Rate Difference = 28.1, 95% CI 2-sided [19.1 to 37.0] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 30.5, 95% CI 2-sided [21.6 to 39.4] — Response Rate Difference = Upadacitinib - Placebo

2. Primary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on DAS28(CRP) at Week 12
Description: The primary endpoint for European Union (EU)/European Medicines Agency (EMA) regulatory purposes was low disease activity, based on a Disease Activity Score 28 (DAS28)-CRP score of ≤ 3.2 at Week 12.
  The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
  A DAS28 score less than or equal to 3.2 indicates low disease activity.
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom DAS28 data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 221 | 221 | 219
percentage of participants | 17.2 [12.2 to 22.2] | 48.4 [41.8 to 55.0] | 47.9 [41.3 to 54.6]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 31.2, 95% CI 2-sided [23.0 to 39.5] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 30.8, 95% CI 2-sided [22.5 to 39.0] — Response Rate Difference = Upadacitinib - Placebo

3. Secondary Outcome: Change From Baseline in in Disease Activity Score 28 (CRP) at Week 12
Description: The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change from Baseline in DAS28 (CRP) indicates improvement in disease activity.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data at Baseline; multiple imputation was used for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 220 | 217 | 219
units on a scale | -1.02 [-1.22 to -0.82] | -2.20 [-2.40 to -2.00] | -2.34 [-2.54 to -2.14]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of covariance (ANCOVA) model with treatment, prior bDMARD use and Baseline value as covariates; Least Squares (LS) Mean Difference = -1.18, 95% CI 2-sided [-1.42 to -0.94] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model with treatment, prior bDMARD use and Baseline value as covariates; LS Mean Difference = -1.32, 95% CI 2-sided [-1.56 to -1.08] — Treatment Difference = Upadacitinib - Placebo

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability.
  A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data at baseline; multiple imputation was used for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 220 | 216 | 219
units on a scale | -0.25 [-0.34 to -0.17] | -0.59 [-0.67 to -0.51] | -0.54 [-0.62 to -0.46]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model with treatment, prior bDMARD use and Baseline value as covariates; LS Mean Difference = -0.33, 95% CI 2-sided [-0.43 to -0.24] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model with treatment, prior bDMARD use and Baseline value as covariates; LS Mean Difference = -0.28, 95% CI 2-sided [-0.38 to -0.18] — Treatment Difference = Upadacitinib - Placebo

5. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Summary (PCS) Score at Week 12
Description: The Short Form 36-Item Health Survey (SF-36) Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component summary score is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The PCS was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from Baseline score indicates an improvement.
Time Frame: Baseline and Week 12
Population: Full analysis set participants with available data; a mixed effect model repeat measurement (MMRM) analysis with data from observed cases to Week 12 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 207 | 209 | 197
units on a scale | 3.03 [1.88 to 4.18] | 7.58 [6.43 to 8.74] | 8.01 [6.84 to 9.18]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; MMRM model with fixed effects of treatment, visit, and treatment-by-visit interaction, previous bDMARD use, and Baseline value as covariate; LS Mean Difference = 4.55, 95% CI 2-sided [3.13 to 5.98] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 4.98, 95% CI 2-sided [3.54 to 6.42] — Treatment Difference = Upadacitinib - Placebo

6. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Based on DAS28 (CRP) at Week 12
Description: Clinical remission (CR) based on DAS28 (CRP) is defined as achieving a DAS28 (CRP) of less than 2.6.
  DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom DAS28 (CRP) data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 221 | 221 | 219
percentage of participants | 10.0 [6.0 to 13.9] | 30.8 [24.7 to 36.9] | 28.3 [22.3 to 34.3]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 20.8, 95% CI 2-sided [13.6 to 28.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 18.4, 95% CI 2-sided [11.2 to 25.5] — Response Rate Difference = Upadacitinib - Placebo

7. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity Based on CDAI at Week 12
Description: Low disease activity based on the clinical disease activity index (CDAI) is defined as a CDAI score ≤ 10.
  CDAI is a composite index for assessing disease activity based on the summation of the total tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity.
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom CDAI data were missing at Week 12 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 221 | 221 | 219
percentage of participants | 19.0 [13.8 to 24.2] | 40.3 [33.8 to 46.7] | 42.0 [35.5 to 48.5]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 21.3, 95% CI 2-sided [13.0 to 29.5] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 23.0, 95% CI 2-sided [14.7 to 31.3] — Response Rate Difference = Upadacitinib - Placebo

8. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Week 12
Description: Participants were asked to indicate the time it took for them to get as limber as possible after awakening with morning stiffness over the past 7 days.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 202 | 207 | 197
minutes | -34.27 [-54.63 to -13.91] | -85.28 [-105.61 to -64.95] | -85.13 [-105.65 to -64.62]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = -51.01, 95% CI 2-sided [-78.14 to -23.87] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = -50.86, 95% CI 2-sided [-78.19 to -23.53] — Treatment Difference = Upadacitinib - Placebo

9. Secondary Outcome: Change From Baseline in in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) at Week 12
Description: The FACIT-Fatigue scale is a 13-item tool that measures an individual's level of fatigue during their usual daily activities over the past 7 days. Each of the fatigue and impact of fatigue items are measured on a five point Likert scale from 0 (not at all) to 4 (very much). The FACIT-Fatigue scale is the sum of the individual 13 scores and ranges from 0 to 52 where higher scores indicate better the quality of life. A positive change from Baseline indicates improvement.
Time Frame: Baseline and week 12
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 207 | 207 | 197
units on a scale | 2.96 [1.62 to 4.30] | 7.91 [6.56 to 9.27] | 7.74 [6.38 to 9.11]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 4.95, 95% CI 2-sided [3.31 to 6.60] — Treatment Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 4.78, 95% CI 2-sided [3.12 to 6.44] — Treatment Difference = Upadacitinib - Placebo

10. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity;
     * Patient global assessment of disease activity;
     * Patient assessment of pain;
     * Health Assessment Questionnaire - Disability Index (HAQ-DI);
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 221 | 221 | 219
percentage of participants | 14.9 [10.2 to 19.6] | 38.0 [31.6 to 44.4] | 43.4 [36.8 to 49.9]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Unadjusted p-value; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 23.1, 95% CI 2-sided [15.1 to 31.0] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Unadjusted p-value; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 28.4, 95% CI 2-sided [20.4 to 36.5] — Response Rate Difference = Upadacitinib - Placebo

11. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR70 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity;
     * Patient global assessment of disease activity;
     * Patient assessment of pain;
     * Health Assessment Questionnaire - Disability Index (HAQ-DI);
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 221 | 221 | 219
percentage of participants | 5.9 [2.8 to 9.0] | 20.8 [15.5 to 26.2] | 26.5 [20.6 to 32.3]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Unadjusted p-value; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 14.9, 95% CI 2-sided [8.7 to 21.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Unadjusted p-value; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 20.6, 95% CI 2-sided [14.0 to 27.2] — Response Rate Difference = Upadacitinib - Placebo

12. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 1
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity;
     * Patient global assessment of disease activity;
     * Patient assessment of pain;
     * Health Assessment Questionnaire - Disability Index (HAQ-DI);
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 1
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 1 or for whom ACR data were missing at Week 1 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 221 | 221 | 219
percentage of participants | 8.6 [4.9 to 12.3] | 22.2 [16.7 to 27.6] | 28.3 [22.3 to 34.3]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Unadjusted p-value; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 13.6, 95% CI 2-sided [7.0 to 20.2] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Unadjusted p-value; [statistical method as in outcome 1, analysis 1]; Response Rate Difference = 19.7, 95% CI 2-sided [12.7 to 26.7] — Response Rate Difference = Upadacitinib - Placebo

ADVERSE EVENTS:
Time Frame: Period 1: From first dose of study drug (placebo or upadacitinib) up to Week 12 or up to 30 days after last dose for participants who discontinued study drug prior to Week 12. Period 1+2: From first dose of upadacitinib up to 30 days after last dose (maximum of 264 weeks).
Groups:
- Period 1: Placebo: Participants received placebo once daily for 12 weeks in Period 1.
- Period 1: Upadacitinib 15 mg: Participants received upadacitinib 15 mg once daily for 12 weeks in Period 1.
- Period 1: Upadacitinib 30 mg: Participants received upadacitinib 30 mg once daily for 12 weeks in Period 1.
- Period 1+2: Upadacitinib 15 mg: Participants originally randomized to upadacitinib 15 mg received upadacitinib 15 mg for 260 weeks and participants originally randomized to placebo followed by upadacitinib 15 mg received upadacitinib 15 mg from Week 12 to Week 260.
- Period1+2: Upadacitinib 30 mg: Participants originally randomized to upadacitinib 30 mg received upadacitinib 30 mg up to Week 260 or implementation of Protocol Amendment 6 (December 2019) and participants originally randomized to placebo followed by upadacitinib 30 mg received upadacitinib 30 mg from Week 12 up to Week 260 or up to implementation of Protocol Amendment 6.
- Period 2: Upadacitinib 15 mg After Switch: Participants who were receiving upadacitinib 30 mg in Period 2 were switched to upadacitinib 15 mg once daily after implementation of Protocol Amendment 6 (December 2019) up to Week 260.
Arm/Group | Period 1: Placebo | Period 1: Upadacitinib 15 mg | Period 1: Upadacitinib 30 mg | Period 1+2: Upadacitinib 15 mg | Period1+2: Upadacitinib 30 mg | Period 2: Upadacitinib 15 mg After Switch
All-Cause Mortality (participants affected / at risk) | 1/221 | 0/221 | 0/219 | 4/324 | 7/321 | 2/179
Serious Adverse Events (participants affected / at risk) | 5/221 | 10/221 | 7/219 | 91/324 | 102/321 | 19/179
Other Adverse Events (participants affected / at risk) | 68/221 | 83/221 | 74/219 | 241/324 | 233/321 | 51/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=221) | Period 1: Upadacitinib 15 mg (N=221) | Period 1: Upadacitinib 30 mg (N=219) | Period 1+2: Upadacitinib 15 mg (N=324) | Period1+2: Upadacitinib 30 mg (N=321) | Period 2: Upadacitinib 15 mg After Switch (N=179)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal decompensation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysbiosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prosthetic cardiac valve stenosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular stent occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 4 (4)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chorioretinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrapulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis B reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster cutaneous disseminated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 11 (13) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salpingo-oophoritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Yersinia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural discharge (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urethral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (11) | 8 (8) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device material issue (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Therapy change (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=221) | Period 1: Upadacitinib 15 mg (N=221) | Period 1: Upadacitinib 30 mg (N=219) | Period 1+2: Upadacitinib 15 mg (N=324) | Period1+2: Upadacitinib 30 mg (N=321) | Period 2: Upadacitinib 15 mg After Switch (N=179)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 20 (24) | 10 (14) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 4 (4) | 17 (26) | 20 (34) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 6 (6) | 13 (21) | 26 (35) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 9 (10) | 5 (5) | 2 (2) | 22 (24) | 15 (15) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 7 (8) | 15 (17) | 3 (3) | 30 (40) | 18 (20) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 2 (2) | 18 (23) | 15 (20) | 1 (2)
BRONCHITIS (Infections and infestations) | 5 (5) | 4 (4) | 5 (5) | 35 (55) | 42 (58) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 20 (21) | 2 (2) | 16 (16)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 27 (29) | 44 (46) | 4 (4)
INFLUENZA (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 15 (18) | 22 (23) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 9 (10) | 12 (13) | 13 (14) | 60 (105) | 45 (75) | 3 (3)
PHARYNGITIS (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 18 (19) | 9 (10) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 6 (6) | 1 (1) | 28 (40) | 22 (23) | 1 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (10) | 12 (12) | 12 (13) | 64 (111) | 57 (84) | 4 (5)
URINARY TRACT INFECTION (Infections and infestations) | 8 (8) | 8 (8) | 6 (6) | 55 (89) | 46 (71) | 4 (4)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (3) | 21 (28) | 17 (19) | 5 (5)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 (5) | 1 (1) | 5 (5) | 36 (42) | 33 (41) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 6 (6) | 2 (2) | 3 (3) | 33 (44) | 25 (31) | 3 (3)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 5 (5) | 7 (7) | 36 (55) | 32 (46) | 1 (1)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 12 (12) | 17 (17) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 23 (28) | 10 (10) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7) | 2 (2) | 31 (37) | 21 (22) | 3 (3)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 10 (11) | 4 (4) | 4 (5) | 36 (54) | 30 (41) | 8 (8)
HEADACHE (Nervous system disorders) | 12 (14) | 9 (9) | 8 (9) | 21 (24) | 21 (24) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (9) | 3 (3) | 24 (28) | 26 (33) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 5 (5) | 6 (7) | 21 (23) | 2 (2)
HYPERTENSION (Vascular disorders) | 4 (4) | 3 (3) | 2 (2) | 41 (45) | 27 (29) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT02675426/Prot_002.pdf
  • Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT02675426/SAP_003.pdf